CLINICAL TRIAL: NCT01901653
Title: Phase I/II Open Label Dose Escalation Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of SC16LD6.5 as a Single Agent in Patients With Recurrent Small Cell Lung Cancer
Brief Title: Rovalpituzumab Tesirine (SC16LD6.5) in Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemcentrx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRX16-001
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Small Cell Lung Cancer
Keywords: Small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rovalpituzumab tesirine (Experimental): Rovalpituzumab tesirine will be administered as a single agent, at increasing dose levels as permitted based on real-time assessment of safety and tolerability, intravenously over 30 minutes. Doses will be repeated on Day 1 of each 21-day or 42-day cycle until either unacceptable toxicity or evidence of disease progression occurs.
  Interventions: Drug: Rovalpituzumab tesirine (SC16LD6.5)

INTERVENTIONS:
Drug: Rovalpituzumab tesirine (SC16LD6.5)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of rovalpituzumab tesirine (SC16LD6.5) at different dose levels in patients with small cell lung cancer whose cancer has progressed or recurred following standard chemotherapy. Once a safe and tolerable dose is determined, the anti-cancer activity of SC16LD6.5 will be assessed by measuring the extent of tumor shrinkage. SC16LD6.5 is an antibody-drug conjugate (ADC). The antibody (SC16) targets a protein that appears to be expressed on the surface of most small cell lung cancers that have been assessed using an immunohistochemical assay. The drug, D6.5, is a very potent form of chemotherapy, specifically a DNA-damaging agent, that is cell cycle independent. ADC's theoretically provide more precise delivery of chemotherapy to cancer cells, possibly improving effectiveness relative to toxicities.

ELIGIBILITY:
Inclusion Criteria

1. Provision of informed consent
2. Male or female ≥18 years of age
3. Histologic or cytologic confirmed diagnosis of small cell lung cancer, either limited or extensive disease at initial presentation is allowed
4. Evidence of progressive disease during or following 1 or 2 prior chemotherapy regimens

   * At least 1 prior regimen must have contained a platinum salt
   * 'Adjuvant therapy' will constitute a prior treatment regimen
   * No more than 2 prior regimens are allowed
5. Measurable disease (only for the phase II portion)
6. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1
7. A minimum life expectancy of 12 weeks
8. Adequate bone marrow, hepatic and renal function as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
   * Serum bilirubin < 1.5 x ULN
   * Aspartate aminotransferase (AST)/Alanine transferase (ALT) (SGOT/SGPT) < 2.5 x ULN for the reference laboratory or < 5 x ULN in the presence of liver metastases
   * Serum creatinine < 1.5 x ULN
9. No 'active' CNS metastases. Prior CNS metastases are allowed, provided adequate palliative therapy has been administered and CNS disease control has been established prior to study entry.

   • A brain MRI scan, ≤ 28 days from day 1, is required
10. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures and who have a negative serum pregnancy test within 1 week prior to initial study treatment. (See Appendix B)
11. Male patients willing to use adequate contraceptive. (See Appendix B)
12. At least 21 days must have elapsed prior to day 1 cycle 1, from chemotherapy, radiotherapy, immunotherapy or following major surgery and any surgical incision should be completely healed. At least 14 days must have elapsed prior to Day 1 Cycle 1 for "limited palliative radiotherapy", defined as a course of therapy encompassing < 25% total bone marrow volume and not exceeding 30 Gy.
13. At least 14 days must have elapsed for chemotherapy regimens, biologic, and targeted therapy given continuously or on a weekly basis with limited potential for delayed toxicity.

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Active involvement of the Central Nervous System (CNS).
3. Uncontrolled infection or systemic disease.
4. Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease e.g. angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
5. Chemotherapy regimens within the last 21 days (or within 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens, biologic, and targeted therapy given continuously or on a weekly basis with limited potential for delayed toxicity within the last 14 days.
6. No concurrent systemic chemotherapy or anticancer biologic therapy is allowed. Note: Patients on hormonal treatment for breast cancer or prostate cancer may continue on treatment and enter into study.
7. Known hypersensitivity to any components of SC16LD6.5 study drug product.
8. Patients with known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both), a history of solid organ or bone marrow transplantation would generally be considered to have met exclusion criteria, however exceptions may be considered on a case-by-case basis by the medical monitor.
9. Psychiatric disorder or social or geographic situation that would preclude study participation.
10. QT interval measurement corrected by Fridericia's formula (QTcF) interval of >450 msec (males) or >470 msec (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Strickland, MD, Study Director — SCRI Innovations
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Blue Ridge Cancer Care, Roanoke, Virginia

REFERENCES:
- [Derived] Rudin CM, Pietanza MC, Bauer TM, Ready N, Morgensztern D, Glisson BS, Byers LA, Johnson ML, Burris HA 3rd, Robert F, Han TH, Bheddah S, Theiss N, Watson S, Mathur D, Vennapusa B, Zayed H, Lally S, Strickland DK, Govindan R, Dylla SJ, Peng SL, Spigel DR; SCRX16-001 investigators. Rovalpituzumab tesirine, a DLL3-targeted antibody-drug conjugate, in recurrent small-cell lung cancer: a first-in-human, first-in-class, open-label, phase 1 study. Lancet Oncol. 2017 Jan;18(1):42-51. doi: 10.1016/S1470-2045(16)30565-4. Epub 2016 Dec 5. PMID 27932068

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1a: Cohort 1 Small Cell Lung Cancer (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.05 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 2 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.1 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 3 (SCLC); Phase 1a: Cohort 8 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.2 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 4 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.4 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 5 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.8 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 6 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.4 mg/kg on Day 1 of every 42-day cycle
- Phase 1a: Cohort 7 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle
- Phase 1a: Cohort 8 Large Cell Neuroendocrine Carcinoma (LCNEC): LCNEC Subjects: Rovalpituzumab tesirine 0.2 mg/kg on Day 1 of every 21-day cycle
- Phase 1b: Retreatment (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles; if eligible, retreatment with rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles. Ongoing subjects from Phase 1a who received an initial dose of 0.2 mg/kg on Day 1 of each 21-day cycle for 3 cycles, and if eligible, retreatment with rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles.
- Phase 1b: Retreatment (LCNEC): LCNEC Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles; if eligible, retreatment with rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles. Ongoing subjects from Phase 1a who received an initial dose of 0.2 mg/kg on Day 1 of each 21-day cycle for 3 cycles, and if eligible, retreatment with rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles.
- Phase 1b: Maintenance (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles; followed by maintenance with rovalpituzumab tesirine 0.1 mg/kg on Day 1 of every 42-day cycle
- Phase 1b: Maintenance (LCNEC): LCNEC Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle for 2 cycles; followed by maintenance with rovalpituzumab tesirine 0.1 mg/kg on Day 1 of every 42-day cycle
Period: Overall Study
Arm/Group | Phase 1a: Cohort 1 Small Cell Lung Cancer (SCLC) | Phase 1a: Cohort 2 (SCLC) | Phase 1a: Cohort 3 (SCLC) | Phase 1a: Cohort 4 (SCLC) | Phase 1a: Cohort 5 (SCLC) | Phase 1a: Cohort 6 (SCLC) | Phase 1a: Cohort 7 (SCLC) | Phase 1a: Cohort 8 (SCLC) | Phase 1a: Cohort 8 Large Cell Neuroendocrine Carcinoma (LCNEC) | Phase 1b: Retreatment (SCLC) | Phase 1b: Retreatment (LCNEC) | Phase 1b: Maintenance (SCLC) | Phase 1b: Maintenance (LCNEC)
Started | 3 | 1 | 11 | 3 | 2 | 3 | 7 | 10 | 1 | 18 | 2 | 16 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 11 | 3 | 2 | 3 | 7 | 10 | 1 | 18 | 2 | 16 | 5
Not completed — Death | 2 | 1 | 8 | 3 | 2 | 2 | 6 | 9 | 1 | 16 | 2 | 15 | 4
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Alive at Study Termination by Sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1a: Cohort 1 (SCLC): SCLC Subjects: Rovalpituzumab tesirine 0.05 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 8 (LCNEC): LCNEC Subjects: Rovalpituzumab tesirine 0.2 mg/kg on Day 1 of every 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Phase 1a: Cohort 1 (SCLC) | Phase 1a: Cohort 2 (SCLC) | Phase 1a: Cohort 3 (SCLC) | Phase 1a: Cohort 4 (SCLC) | Phase 1a: Cohort 5 (SCLC) | Phase 1a: Cohort 6 (SCLC) | Phase 1a: Cohort 7 (SCLC) | Phase 1a: Cohort 8 (SCLC) | Phase 1a: Cohort 8 (LCNEC) | Phase 1b: Retreatment (SCLC) | Phase 1b: Retreatment (LCNEC) | Phase 1b: Maintenance (SCLC) | Phase 1b: Maintenance (LCNEC) | Total
Number analyzed (Participants) | 3 | 1 | 11 | 3 | 2 | 3 | 7 | 10 | 1 | 18 | 2 | 16 | 5 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 6 | 2 | 2 | 1 | 5 | 7 | 1 | 11 | 1 | 9 | 2 | 51
  >=65 years | 0 | 0 | 5 | 1 | 0 | 2 | 2 | 3 | 0 | 7 | 1 | 7 | 3 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 2 | 1 | 1 | 2 | 4 | 0 | 11 | 0 | 4 | 2 | 34
  Male | 1 | 0 | 7 | 1 | 1 | 2 | 5 | 6 | 1 | 7 | 2 | 12 | 3 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 1 | 10 | 3 | 2 | 3 | 7 | 10 | 1 | 14 | 2 | 15 | 4 | 75
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 3 | 1 | 10 | 2 | 2 | 2 | 5 | 10 | 1 | 15 | 2 | 15 | 3 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 11 | 3 | 2 | 3 | 7 | 10 | 1 | 18 | 2 | 16 | 5 | 82
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOGScale:Score-Description:0-Normalactivity.Fullyactive,abletocarryonallprediseaseperformancew/orestriction/1-Symptoms,but ambulatory.Restrictedinphysicallystrenuousactivity,butambulatoryandabletocarryoutworkofa light/sedentarynature(eg,light housework,office work)/2-In bed<50%ofthetime.Ambulatoryandcapableofallselfcare,but unabletocarryoutanyworkactivities.Upandabout>50%ofwakinghours/3-In bed>50%ofthetime.Capableofonlylimitedselfcare,confinedtobed/chair>50%ofwakinghours/4-100% bedridden.Completelydisabled.Cannotcarryonanyselfcare.Totallyconfinedtobed/chair/5-Dead.
  Participants
    0 | 2 | 0 | 4 | 2 | 1 | 1 | 0 | 3 | 0 | 3 | 1 | 5 | 1 | 23
    1 | 1 | 1 | 7 | 1 | 1 | 2 | 6 | 7 | 1 | 13 | 1 | 11 | 3 | 55
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Rovalpituzumab Tesirine
Description: MTD was determined by testing increasing doses from 0.05 mg/kg up to 0.8 mg/kg on Day 1 of every 21-day or 42-day cycle, Phase 1a cohorts 1 to 8. MTD will be defined as the dose level immediately below the dose level at which ≥ 2 of the first 3 subjects per cohort (or ≥ 2 of 6 subjects) during the first cycle experience a study drug related dose limiting toxicity (DLT).
Time Frame: The DLT period was defined as either 21 or 42 days following the first dose of Rovalpituzumab tesirine during dose escalation (Phase 1a), depending on Cycle length.
Population: All subjects from Phase 1a Dose Escalation: Cohort 1 to 8 who received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- Rovalpituzumab Tesirine: Rovalpituzumab tesirine (SC16LD6.5) will be administered intravenously (IV) to subjects with recurrent small cell lung cancer. Rovalpituzumab tesirine will be given on Day 1 of every 21-day or 42-day cycle.
Arm/Group | Rovalpituzumab Tesirine
Number analyzed (Participants) | 41
mg/kg | 0.4

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Overall response was assessed at each visit post-baseline based on a subject's lesion measurements or assessments (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD], or not evaluable as defined by RECIST v1.1, plus an additional category of early death). The best overall response was then determined. A subject was defined as having an objective response if they had a best overall response of CR or PR prior to receiving any subsequent anticancer therapy; confirmed response is confirmation of CR or PR at least 4 weeks from the initial determination per RECIST v1.1. Subjects with a post-baseline assessment were included in the calculations for objective response rate (ORR).
  Outcome is based on data reported by Investigator (INV); available and evaluable radiographic scans were collected retrospectively for review by an Independent Review Committee (IRC).
Time Frame: From first dose of rovalpituzumab tesirine to last event, up through study completion (on average approximately 4 months).
Population: Subjects with at least one post-dose assessment. All LCNEC subjects were analyzed. No LCNEC subjects achieved CR or PR and, therefore, the ORR was 0%.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- SCLC Subjects: SCLC Subjects who received rovalpituzumab tesirine 0.2 mg/kg to 0.4 mg/kg
- LCNEC Subjects: LCNEC Subjects who received rovalpituzumab tesirine 0.2 mg/kg to 0.4 mg/kg
Arm/Group | SCLC Subjects | LCNEC Subjects
Number analyzed (Participants) | 67 | 8
percentage of subjects
  ORR unconfirmed by Investigator | 25 [14.98 to 38.44] | 0 [0 to 36.94]
  ORR confirmed by Investigator | 17 [8.44 to 28.97] | 0 [0 to 36.94]
  ORR unconfirmed by IRC | 27 [16.14 to 40.96] | 0 [0 to 39.94]
  ORR confirmed by IRC | 16 [7.77 to 28.8] | 0 [0 to 36.94]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as the number of months from the initial CR or PR to the time of disease progression or death, whichever occurred first.
  Outcome is based on data reported by Investigator (INV); available and evaluable radiographic scans were collected retrospectively for review by an Independent Review Committee (IRC).
Time Frame: From first dose of Rovalpituzumab tesirine to last event timepoint, up through study completion (on average approximately 4 months, but up to 6.51 months).
Population: Subjects with at least one post-dose assessment. No LCNEC subjects achieved CR or PR, therefore DOR was not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SCLC Subjects | LCNEC Subjects
Number analyzed (Participants) | 67 | 0
months
  DOR by INV | 2.89 [2.17 to 6.51] |
  DOR by IRC | 1.71 [0.03 to 3.06] |

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit is defined as a subject with best Overall Response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) prior to receiving any subsequent anticancer therapy; as defined by RECIST version 1.1. CBR is defined as the proportion of subjects with Clinical Benefit based on assessment of overall response. CBR will be presented as a number and percentage with 95% confidence bounds. Any subjects not exhibiting a response (CR or PR or SD) are considered non-responders.
  Outcome is based on data reported by Investigator (INV); available and evaluable radiographic scans were collected retrospectively for review by an Independent Review Committee (IRC).
Time Frame: From first dose of Rovalpituzumab tesirine to last event timepoint, up through study completion (on avergae approximately 4 months).
Population: Subjects with at least one post-dose assessment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | SCLC Subjects | LCNEC Subjects
Number analyzed (Participants) | 67 | 8
percentage of subjects
  CBR unconfirmed by INV | 73 [59.73 to 83.64] | 88 [47.35 to 99.68]
  CBR confirmed by INV | 58 [44.07 to 70.39] | 75 [34.91 to 96.81]
  CBR unconfirmed by IRC | 75 [61 to 85.33] | 75 [34.91 to 96.81]
  CBR confirmed by IRC | 56 [42.32 to 69.7] | 75 [34.91 to 96.81]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the number of months from the first day of study drug administration to disease recurrence or progression, or death on study.
  Outcome is based on data reported by Investigator (INV); available and evaluable radiographic scans were collected retrospectively for review by an Independent Review Committee (IRC).
Time Frame: From first dose of rovalpituzumab tesirine to last event timepoint, up through study completion (approximately 4 months on average, but up to 14.46 months).
Population: Subjects with at least one post-dose assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SCLC Subjects | LCNEC Subjects
Number analyzed (Participants) | 67 | 8
months
  PFS by INV | 2.79 [2.33 to 3.71] | 3.07 [1.45 to 6.83]
  PFS by IRC | 2.89 [2.14 to 3.84] | 2.6 [1.25 to 14.46]

6. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the first day of study treatment to death. Subjects who were alive were censored at the date of last known alive.
Time Frame: From first dose of Rovalpituzumab tesirine to last event, up through study completion (on average approximately 5-7 months, but up to 14.6 months).
Population: Subjects with at least one post-dose assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SCLC Subjects | LCNEC Subjects
Number analyzed (Participants) | 67 | 8
months | 4.76 [4.01 to 7.13] | 6.59 [2.89 to 14.46]

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of Rovalpituzumab Tesirine Antibody Drug Conjugate (ADC)
Description: The maximum serum concentration (Cmax; measured in μg/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing cycle.
Time Frame: From Day 1 of first dose to End of Dose Cycle
Population: All subjects who received at least 1 dose of study drug, with evaluable data at each given timepoint. For Phase 1b, pharmacokinetic (PK) sampling was sparse; therefore, pharmacokinetic parameters were not estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Phase 1a: Cohort 1: All Subjects: Rovalpituzumab tesirine 0.05 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 2: All Subjects: Rovalpituzumab tesirine 0.1 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 3; Phase 1a: Cohort 8: All Subjects: Rovalpituzumab tesirine 0.2 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 4: All Subjects: Rovalpituzumab tesirine 0.4 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 5: All Subjects: Rovalpituzumab tesirine 0.8 mg/kg on Day 1 of every 21-day cycle
- Phase 1a: Cohort 6: All Subjects: Rovalpituzumab tesirine 0.4 mg/kg on Day 1 of every 42-day cycle
- Phase 1a: Cohort 7: All Subjects: Rovalpituzumab tesirine 0.3 mg/kg on Day 1 of every 42-day cycle
Arm/Group | Phase 1a: Cohort 1 | Phase 1a: Cohort 2 | Phase 1a: Cohort 3 | Phase 1a: Cohort 4 | Phase 1a: Cohort 5 | Phase 1a: Cohort 6 | Phase 1a: Cohort 7 | Phase 1a: Cohort 8
Number analyzed (Participants) | 3 | 1 | 10 | 3 | 2 | 3 | 10 | 11
μg/mL | 1.27 (13) | 2.42 | 5.08 (21) | 8.81 (7) | 18.8 (27) | 11.4 (27) | 7.67 (21) | 5.36 (26)

8. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC) of Rovalpituzumab Tesirine ADC
Description: The area under the serum concentration-time curve (AUC; measured in μg•d/mL) is a method of measurement to determine the total exposure of a drug in blood serum.
Time Frame: From Day 1 of first dose to End of Dose Cycle
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•d/mL
Arm/Group | Phase 1a: Cohort 1 | Phase 1a: Cohort 2 | Phase 1a: Cohort 3 | Phase 1a: Cohort 4 | Phase 1a: Cohort 5 | Phase 1a: Cohort 6 | Phase 1a: Cohort 7 | Phase 1a: Cohort 8
Number analyzed (Participants) | 3 | 1 | 10 | 3 | 2 | 3 | 10 | 11
μg•d/mL | 12.3 (22) | 26.3 | 45.6 (32) | 97.3 (21) | 142 (18) | 107 (28) | 64.8 (36) | 45.0 (34)

ADVERSE EVENTS:
Time Frame: From date of first dose through 30-days following last dose (on average 85 days).
Arm/Group | Phase 1a: Cohort 1 (SCLC) | Phase 1a: Cohort 2 (SCLC) | Phase 1a: Cohort 3 (SCLC) | Phase 1a: Cohort 4 (SCLC) | Phase 1a: Cohort 5 (SCLC) | Phase 1a: Cohort 6 (SCLC) | Phase 1a: Cohort 7 (SCLC) | Phase 1a: Cohort 8 (SCLC) | Phase 1a: Cohort 8 (LCNEC) | Phase 1b: Retreatment (SCLC) | Phase 1b: Retreatment (LCNEC) | Phase 1b: Maintenance (SCLC) | Phase 1b: Maintenance (LCNEC)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 3/11 | 3/3 | 2/2 | 2/3 | 1/7 | 4/10 | 1/1 | 7/18 | 1/2 | 5/16 | 4/5
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 11/11 | 3/3 | 2/2 | 3/3 | 7/7 | 10/10 | 1/1 | 18/18 | 2/2 | 15/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: Cohort 1 (SCLC) (N=3) | Phase 1a: Cohort 2 (SCLC) (N=1) | Phase 1a: Cohort 3 (SCLC) (N=11) | Phase 1a: Cohort 4 (SCLC) (N=3) | Phase 1a: Cohort 5 (SCLC) (N=2) | Phase 1a: Cohort 6 (SCLC) (N=3) | Phase 1a: Cohort 7 (SCLC) (N=7) | Phase 1a: Cohort 8 (SCLC) (N=10) | Phase 1a: Cohort 8 (LCNEC) (N=1) | Phase 1b: Retreatment (SCLC) (N=18) | Phase 1b: Retreatment (LCNEC) (N=2) | Phase 1b: Maintenance (SCLC) (N=16) | Phase 1b: Maintenance (LCNEC) (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cauda Equina Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Capillary Leak Syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: Cohort 1 (SCLC) (N=3) | Phase 1a: Cohort 2 (SCLC) (N=1) | Phase 1a: Cohort 3 (SCLC) (N=11) | Phase 1a: Cohort 4 (SCLC) (N=3) | Phase 1a: Cohort 5 (SCLC) (N=2) | Phase 1a: Cohort 6 (SCLC) (N=3) | Phase 1a: Cohort 7 (SCLC) (N=7) | Phase 1a: Cohort 8 (SCLC) (N=10) | Phase 1a: Cohort 8 (LCNEC) (N=1) | Phase 1b: Retreatment (SCLC) (N=18) | Phase 1b: Retreatment (LCNEC) (N=2) | Phase 1b: Maintenance (SCLC) (N=16) | Phase 1b: Maintenance (LCNEC) (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4 | 0 | 5 | 1 | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 3 | 0 | 4 | 2
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 0
Periorbital Oedema (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 0 | 1 | 4 | 0 | 8 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 8 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 2 | 0 | 2 | 2 | 0 | 4 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 3 | 2 | 2 | 3 | 2 | 6 | 0 | 12 | 1 | 5 | 5
Oedema Peripheral (General disorders) | 2 | 0 | 4 | 0 | 0 | 2 | 1 | 2 | 0 | 7 | 1 | 6 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 4 | 1
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 0
Face Oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Lipase Increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2
Amylase Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Weight Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1 | 2 | 3 | 0 | 1 | 4 | 0 | 6 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 1 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 1 | 7 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 1 | 10 | 1 | 4 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 0 | 2 | 2 | 2 | 0 | 3 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 3 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 6 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.